CLINICAL TRIAL: NCT03726528
Title: Optimized Characterization of Takotsubo Syndrome by Obtaining Pressure Volume Loops
Acronym: OCTOPUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Ingo Eitel, MD, Director, University of Luebeck
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-078
Record Dates: First submitted 2018-10-01; First posted 2018-10-31 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Takotsubo Syndrome
MeSH Terms: conditions — Takotsubo Cardiomyopathy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental intervention (Experimental)
  Interventions: Diagnostic Test: Measurements of left ventricular pressure and volume

INTERVENTIONS:
Diagnostic Test: Measurements of left ventricular pressure and volume — Patients with suspected Takotsubo syndrome (typical ballooning in left ventriculography without significant obstructive coronary artery disease that sufficiently explains the contraction abnormalities) will undergo continuous online measurements of left ventricular pressure and volume using conductance catheters. Cardiac magnetic resonance (CMR) imaging will be performed in patients without contraindications for optimized morphological characterization and exclusion of important differential diagnoses.

SUMMARY:
Aim of this prospective study is to assess the pathophysiology of Takotsubo Syndrome by obtaining pressure volume loops with conductance catheters, which allows detailed conclusions regarding systolic and diastolic hemondynamics and subsequently regarding potential underlying mechanisms

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Takotsubo syndrome according to current diagnostic criteria including complete normalization of left ventricular function during follow-up
* Sinus rhythm during invasive measurements
* Age ≥18 years
* Written informed consent

Exclusion Criteria:

* Cardiogenic shock
* Signs of myocarditis or myocardial infarction with spontaneous lysis of thrombus in cardiac magnetic resonance imaging
* Pregnancy
* Participation in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Changes in contractility derived from pressure-volume measurements | Day 0
  systolic/diastolic pressure-volume relationship (mmHg/ml)
Changes in contractility derived from pressure-volume measurements | Day 0
  peak-power index (mmHG/s)
Changes in contractility derived from pressure-volume measurements | Day 0
  peak filling rate (ml/s)
Changes in contractility derived from pressure-volume measurements | Day 0
  stroke work (mmHG x ml)
Changes in contractility derived from pressure-volume measurements | Day 0
  relaxation constant "Tau" (ms)
Changes in contractility derived from pressure-volume measurements | Day 0
  time to Emax (ms)
Changes in contractility derived from pressure-volume measurements | Day 0
  max/min rate of left ventricular pressure change (mmHg/s)

SECONDARY OUTCOMES:
Energetic parameters derived from pressure-volume measurements | Day 0
  stroke work, potential energy (mmHg x ml)
Energetic parameters derived from pressure-volume measurements | Day 0
  total pressure volume area (mmHg/ml)
Afterload parameters derived from pressure-volume measurements | Day 0
  arterial elastance (mmHg/ml)
Afterload parameters derived from pressure-volume measurements | Day 0
  ventricular arterial coupling (no dimension)
Afterload parameters derived from pressure-volume measurements | Day 0
  total arterial compliance (mmHg/ml)
- Correlation of pressure-volume measurements with morphological and functional findings in CMR imaging | Day 3
  (presence of myocardial edema or late gadolinium enhancement, native T1 time, myocardial strain assessed by CMR feature tracking)
- Correlation of pressure-volume measurements with biomarker release | Day 0
  (troponin, NT-proBNP)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical clinic II-UKSH, Lübeck, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Stiermaier T, Reil JC, Sequeira V, Rawish E, Mezger M, Patz T, Paitazoglou C, Schmidt T, Frerker C, Steendijk P, Reil GH, Eitel I. Hemodynamic Assessment in Takotsubo Syndrome. J Am Coll Cardiol. 2023 May 23;81(20):1979-1991. doi: 10.1016/j.jacc.2023.03.398. PMID 37197841